CLINICAL TRIAL: NCT01504854
Title: Phase II Study to Evaluate the Impact on Biomarkers of Resveratrol Treatment in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Resveratrol for Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADC-037-RES
Record Dates: First submitted 2011-12-23; First posted 2012-01-06 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Dementia; Brain diseases; Resveratrol; Memory problems; Mental disorders; Cognitive disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Memory Disorders; Mental Disorders; Cognitive Dysfunction | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resveratrol (Experimental): Subjects will take 500 mg by mouth once daily increasing at 13 week intervals to a maximum of 1 gram by mouth twice daily with or without food.
  Interventions: Drug: Resveratrol
- Placebo (Placebo Comparator): Subjects will receive a matching placebo to be taken with or without food.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Resveratrol — The dosage will begin at 500 mg taken once daily and increase at 13 week intervals to 1 gram taken by mouth twice daily, supplied as 500 mg capsules (two capsules twice daily).
  Arms: Resveratrol
Drug: Placebo — The matching placebo will begin at a capsule taken once daily and increase at 13 week intervals to two capsules twice daily.
  Arms: Placebo

SUMMARY:
Resveratrol is derived from plants and is found in highest levels in red wine and the skin of red grapes. A recent study reported that monthly and weekly consumption of red wine is associated with a lower risk of dementia. There is compelling evidence that caloric restriction can improve overall health by activating a class of enzymes known as Sirtuins. Resveratrol is a substance found in some plants that directly activates sirtuins, mimicking the effects of caloric restriction and may affect regulatory pathways of diseases of aging, including Alzheimer's disease (AD).

In this study, people with AD will be given either Resveratrol or placebo for 12 months to determine whether daily resveratrol therapy is beneficial in delaying or altering the deterioration of memory and daily functioning. Subjects age 50 and above with a diagnosis of probable AD may qualify for participation in this study. A small group of 15 participants will be asked to take part in a more detailed 24-hour Pharmacokinetic (PK) sub-study that will measure resveratrol levels over a 24 hour period.

DETAILED DESCRIPTION:
This double blind, placebo-controlled trial will be conducted at approximately 26 Alzheimer's Disease Cooperative Study (ADCS) clinical centers. One hundred twenty (120) patients with mild to moderate dementia due to probable Alzheimer's disease (AD) will be randomly assigned to treatment (1:1) with resveratrol starting at 500 mg once daily or matching placebo, increasing at 13 week intervals to a maximum of 1 gram twice daily (divided into two 500 mg capsules taken orally) taken with or without food. Participants will be treated for 52 weeks, and will undergo venous blood draws for biomarker analysis at Baseline and at 52 weeks; participants will also undergo two lumbar punctures for biomarker analyses of cerebrospinal fluid (CSF) at Baseline and at Week 52. Participants will undergo magnetic resonance imaging (MRI) to measure rate of whole-brain and regional atrophy at Screening, Week 13 and Week 52 visits. Randomization will be stratified by site. For monitoring of potential toxicities of the study drug - particularly nephrotoxicity - subjects will undergo physical examination, neurological examination, adverse event review, blood chemistries to include blood urea nitrogen (BUN) and Creatinine (Cr), pharmacokinetic (PK) analyses for resveratrol and its metabolites, and urinalysis every 6-7 weeks during the study. Clinical, Cognitive and Functional effects of resveratrol and insulin and glucose metabolism will also be assessed.

A subgroup of approximately 15 subjects enrolled will be randomized 4:1 (N = 15, 12 treated + 3 placebo) for more detailed 24-hour PK analysis. For these individuals, blood samples will be collected at 15 different time points. Measurements will include levels of resveratrol and its major metabolites (sulfated- and glucuronidated-resveratrol). These subjects will complete the detailed PK with each dosage step. This 24-hour PK sampling in the subgroup will occur after the first dose following Baseline, after the first dose at each dose increment (Weeks 13, 26 and 39), and after the final dose (Week 52).

Enrollment will be restricted to individuals who are able to abstain from ingesting large quantities of resveratrol-containing foods (including red wine). 1-2 glasses of red wine or red grape juice and 1 serving of red grapes daily is acceptable. Subjects must also be able to abstain from ingesting herbal/natural preparations or dietary supplements containing resveratrol.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD (NINDS-ADRDA criteria).
* Age must be 50 years or older.
* Able to ingest oral medications.
* Caregiver/Study Partner who has direct contact with the participant more than 2 days per week to accompany participant to all visits.
* MMSE score between 14 and 26 (inclusive).
* Modified Hachinski score of less than or equal to 4.
* Able to abstain from ingesting large quantities of resveratrol-containing foods (including red wine). 1-2 glasses of red wine or red grape juice daily acceptable; 1 serving of red grapes daily acceptable.
* Able to abstain from ingesting herbal/natural preparations or dietary supplements containing resveratrol.

Exclusion Criteria:

* Non-AD dementia.
* Probable AD with Down syndrome.
* History of clinically significant stroke.
* Current evidence or history in past two years of epilepsy, focal brain lesion, head injury with loss of consciousness or DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse.
* Sensory impairment that would preclude the participant from participating in or cooperating with the protocol.
* Use of investigational agent within two months of Screening.
* Evidence of any significant clinical disorder or laboratory finding that renders the participant unsuitable for receiving an investigational drug including clinically significant or unstable hematologic, hepatic, cardiovascular, pulmonary, gastrointestinal, endocrine, metabolic, renal or other systemic disease or laboratory abnormality.
* Active neoplastic disease, history of cancer five years prior to screening, including breast cancer (history or skin melanoma or stable prostate cancer are not excluded).
* History of seizure within past five years.
* Pregnancy or possible pregnancy.
* Use of resveratrol containing supplements.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond S. Turner, MD, PhD, Study Director — Georgetown University
Locations (26):
- United States (26):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - University of California, Irvine, Irvine, California
  - University of California, San Diego - Comprehensive Alzheimer's Program, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - New York University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Case Western Reserve University, Beachwood, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, North Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - U of WA / VA Puget Sound Alzheimer's Disease Research Center, Seattle, Washington

REFERENCES:
- [Background] Vang O, Ahmad N, Baile CA, Baur JA, Brown K, Csiszar A, Das DK, Delmas D, Gottfried C, Lin HY, Ma QY, Mukhopadhyay P, Nalini N, Pezzuto JM, Richard T, Shukla Y, Surh YJ, Szekeres T, Szkudelski T, Walle T, Wu JM. What is new for an old molecule? Systematic review and recommendations on the use of resveratrol. PLoS One. 2011;6(6):e19881. doi: 10.1371/journal.pone.0019881. Epub 2011 Jun 16. PMID 21698226
- [Background] Smoliga JM, Baur JA, Hausenblas HA. Resveratrol and health--a comprehensive review of human clinical trials. Mol Nutr Food Res. 2011 Aug;55(8):1129-41. doi: 10.1002/mnfr.201100143. Epub 2011 Jun 20. PMID 21688389
- [Background] Patel KR, Scott E, Brown VA, Gescher AJ, Steward WP, Brown K. Clinical trials of resveratrol. Ann N Y Acad Sci. 2011 Jan;1215:161-9. doi: 10.1111/j.1749-6632.2010.05853.x. PMID 21261655
- [Background] Timmers S, Konings E, Bilet L, Houtkooper RH, van de Weijer T, Goossens GH, Hoeks J, van der Krieken S, Ryu D, Kersten S, Moonen-Kornips E, Hesselink MKC, Kunz I, Schrauwen-Hinderling VB, Blaak E, Auwerx J, Schrauwen P. Calorie restriction-like effects of 30 days of resveratrol supplementation on energy metabolism and metabolic profile in obese humans. Cell Metab. 2011 Nov 2;14(5):612-22. doi: 10.1016/j.cmet.2011.10.002. PMID 22055504
- [Background] Albani D, Polito L, Forloni G. Sirtuins as novel targets for Alzheimer's disease and other neurodegenerative disorders: experimental and genetic evidence. J Alzheimers Dis. 2010;19(1):11-26. doi: 10.3233/JAD-2010-1215. PMID 20061622
- [Derived] Greco GA, Rock M, Amontree M, Lanfranco MF, Korthas H, Hong SH, Turner RS, Rebeck GW, Conant K. CCR5 deficiency normalizes TIMP levels, working memory, and gamma oscillation power in APOE4 targeted replacement mice. Neurobiol Dis. 2023 Apr;179:106057. doi: 10.1016/j.nbd.2023.106057. Epub 2023 Mar 5. PMID 36878326
- [Derived] Stites SD, Turner RS, Gill J, Gurian A, Karlawish J, Grill JD; Alzheimer's Disease Cooperative Study. Research Attitudes Questionnaire scores predict Alzheimer's disease clinical trial dropout. Clin Trials. 2021 Apr;18(2):237-244. doi: 10.1177/1740774520982315. Epub 2021 Jan 10. PMID 33426901
- [Derived] Moussa C, Hebron M, Huang X, Ahn J, Rissman RA, Aisen PS, Turner RS. Resveratrol regulates neuro-inflammation and induces adaptive immunity in Alzheimer's disease. J Neuroinflammation. 2017 Jan 3;14(1):1. doi: 10.1186/s12974-016-0779-0. PMID 28086917
- See also: Alzheimer's Disease Cooperative Study — http://adcs.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multicenter, double-blind, placebo-controlled trial was conducted June 2012-March 2014 with participants recruited from 26 US academic clinics affiliated with the Alzheimer's Disease Cooperative Study (ADCS).
Pre-assignment Details: 119 subjects were recruited rather than 120.
Period: Overall Study
Arm/Group | Resveratrol | Placebo
Started | 64 | 55
Completed | 56 | 48
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Resveratrol: 60 subjects will take 500 mg by mouth once daily increasing at 13 week intervals to a maximum of 1 gram by mouth twice daily with or without food.
  Resveratrol: The dosage will begin at 500 mg taken once daily and increase at 13 week intervals to 1 gram taken by mouth twice daily, supplied as 500 mg capsules (two capsules twice daily).
- Placebo: 60 subjects will receive a matching placebo to be taken with or without food.
  Placebo: The matching placebo will begin at a capsule taken once daily and increase at 13 week intervals to two capsules twice daily.
- Total: Total of all reporting groups
Arm/Group | Resveratrol | Placebo | Total
Number analyzed (Participants) | 64 | 55 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (7.7) | 73 (8.2) | 71.4 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 28 | 68
  Male | 24 | 27 | 51

OUTCOME MEASURES:

1. Post Hoc Outcome: Change From Baseline in Cerebrospinal Fluid Amyloid β40 Concentration at 52 Weeks
Description: Mean change from baseline in cerebrospinal fluid amyloid β40 concentration at 52 weeks
Time Frame: Baseline and Week 52
Population: Post-hoc modified intention-to-treat (ITT) re-analysis of primary outcomes at Week 52 adjusting for age and AD duration in the mixed-model repeated measures model
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 56 | 48
ng/ml | 6456 (2282) | 5622 (1736)

2. Primary Outcome: Number of Adverse Events
Description: The safety and tolerability of treatment with resveratrol will be assessed by analysis of adverse events, including symptoms, abnormal findings on physical examinations, standard laboratory tests and PK analysis of resveratrol and its major metabolites. The frequencies of adverse events or laboratory abnormalities between the participants who receive resveratrol and those receiving placebo will be compared.
Time Frame: Baseline, Weeks 6, 13, 19, 26, 32, 39, 45, and 52
Population: ITT population
Measure: Number; unit: number of AEs
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 56 | 48
number of AEs | 355 | 302

3. Primary Outcome: Change From Baseline in Volumetric Magnetic Resonance Imaging (MRI)
Description: MRI will be used to assess the effect of treatment on rate of whole brain volume
Time Frame: Baseline and Week 52
Population: ITT population
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 56 | 48
cm^3 | 27 (12) | 10 (7)

4. Secondary Outcome: Change in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL)
Description: The ADCS-ADL is an activities of daily living inventory developed by the ADCS to assess functional performance in participants with AD. The ADCS-ADL includes some items from traditional basic ADL tests (e.g., grooming, dressing, walking, bathing, feeding, toileting) as well as instrumental (complex) activities of daily living (e.g., shopping, preparing meals, using household appliances, keeping appointments, reading). This structured questionnaire is administered to the subject's caregiver/study partner. The range of this instrument is 0 to 78 with lower numbers indicating greater impairment.
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 56 | 48
units on a scale | 6.3 (11.6) | 9.2 (12.6)

5. Secondary Outcome: Comparison of the Response to Treatment of Resveratrol Based on ApoE Genotype
Description: CSF Abeta40
Time Frame: Week 52
Population: ITT analyses. Total population and subpopulation of ApoE4 non-carriers.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 56 | 48
ng/ml
  Total Population | 6574 (2346) | 6560 (2190)
  ApoE4 non-carriers | 5859 (2085) | 6339 (1709)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 52 week period (the duration of the subject's participation in the study).
Description: Participants received physical and neurologic examinations and vital signs at each visit. Site investigators classified AEs by severity and causality. If a participant withdrew, an early termination visit similar to a baseline visit was scheduled. An independent Data and Safety Monitoring Board reviewed data quarterly.
Arm/Group | Resveratrol | Placebo
Serious Adverse Events (participants affected / at risk) | 13/64 | 10/55
Other Adverse Events (participants affected / at risk) | 64/64 | 52/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resveratrol (N=64) | Placebo (N=55)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Subdural hematoma (Nervous system disorders) | 0 (0) | 1 (1)
Unresponsiveness (Nervous system disorders) | 0 (0) | 1 (1)
Altered mental state (Nervous system disorders) | 1 (1) | 0 (0)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
"Blood clots" in the lung/pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Melanoma of the lung, Stage 4 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large pleural effusion secondary to stage 4 melanoma of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Syncope/atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Infections (Infections and infestations) | 0 (0) | 1 (1)
Rhabdomyolosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Low hemoglobin (Investigations) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Drowning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Left femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complications from colostomy reversal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Water intoxication (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Altered mental state (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 1 (1)
Perforated viscus with perforated sigmoid diverticulitis with peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Right peripheral vascular disease (status post Carotid Endarterectomy) (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resveratrol (N=64) | Placebo (N=55)
Diarrhoea (Gastrointestinal disorders) | 26 (26) | 7 (7)
Urinary Tract Infection (Infections and infestations) | 19 (19) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 22 (22) | 14 (14)
Dizzyness (Nervous system disorders) | 6 (6) | 5 (5)
Headache (Nervous system disorders) | 11 (11) | 6 (6)
Anxiety (Psychiatric disorders) | 3 (3) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (7)
Hypertension (Vascular disorders) | 4 (4) | 3 (3)

LIMITATIONS AND CAVEATS:
This phase 2 study has limitations. A larger study is required to determine whether resveratrol may be beneficial. More potent and bioavailable SIRT1 activators are also in development.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No